CLINICAL TRIAL: NCT00274222
Title: The Role of Nebulized Budesonide in the Treatment of Acute Exacerbations of COPD
Status: Terminated | Type: Observational
Sponsor: Inonu University (Other)
Other Study IDs: 2006-3
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2006-01-10 (Estimated); Status verified 2006-01

CONDITIONS: COPD Acute Exacerbation
Keywords: COPD, nebulized budesonide, systemic corticosteroids
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

SUMMARY:
This study was designed to evaluate the hypothesis that nebulized budesonide) might be an alternative to systemic corticosteroids (SC) in the treatment of patients with acute exacerbations of COPD (AECOPD).

DETAILED DESCRIPTION:
Patients, hospitalized with AECOPD, were randomized into three groups. Group I received only bronchodilator treatment (BDT), Group II received SC (40 mg prednisolon) plus BDT, and Group III received nebulized budesonide (NB)(1500 mcg qid) plus BDT. Improvement rates in multiple parameters during 10-day hospitalization, and acute exacerbation and re-hospitalization rates within one-month after discharge were compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients who were admitted to our pulmonary department for an acute exacerbation were prospectively enrolled in the study

Exclusion Criteria:

* COPD patients hospitalized with specific reasons like pneumonia, pulmonary emboli, congestive heart failure, pneumothorax etc. as the cause of acute exacerbation, or patients with risk of imminent respiratory failure requiring mechanical ventilation or direct admission to the ICU were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-01; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: HAKAN GUNEN, MD, Study Chair — INONU UNIVERSITY PULMONARY MEDICINE